CLINICAL TRIAL: NCT05397496
Title: A Phase I, Open-label, Multi-center Study of PIT565 in Patients With Relapsed and/or Refractory B-cell Malignancies
Brief Title: Study of PIT565 in Relapsed and/or Refractory B-cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPIT565A12101; 2022-000367-45 (EudraCT Number)
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: B-cell Non-Hodgkin Lymphoma (B-NHL); B-cell Acute Lymphoblastic Leukemia (B-ALL)
Keywords: Phase I; Trispecific antibody; Non-Hodgkin lymphoma; Acute Lymphoblastic Leukemia; PIT565
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PIT565 Group A (dose escalation part) (Experimental): PIT565 in adult NHL patients for whom two or more lines of chemotherapy have failed and either having progressed (or relapsed) after autologous hematopoietic stem cell transplantation (HSCT), or being ineligible for or not consenting to the procedure
  Interventions: Biological: PIT565
- PIT565 Group B (dose escalation part) (Experimental): PIT565 in adult R/R ALL patients
  Interventions: Biological: PIT565
- PIT565 Group A1 (dose expansion part) (Experimental): PIT565 Recommended dose 1 (RD1) in adult R/R large B-cell lymphoma (LBCL) (DLBCL, double/triple hit High-grade B-cell lymphoma (HGBCL), Primary mediastinal large B-cell lymphoma (PMBCL), Follicular lymphoma grade 3B (FL3B)) patients
  Interventions: Biological: PIT565
- PIT565 Group A2 (dose expansion part) (Experimental): PIT565 RD2 in adult R/R LBCL (DLBCL, double/triple hit HGBCL, PMBCL, FL3B) patients
  Interventions: Biological: PIT565
- PIT565 Group B1 (dose expansion part) (Experimental): PIT565 in adult R/R ALL patients
  Interventions: Biological: PIT565

INTERVENTIONS:
Biological: PIT565 — Intravenous (i.v.) infusion or Subcutaneous (s.c.) injection

SUMMARY:
This is an open-label, multicenter, phase I study, which primary objective is to characterize the safety and tolerability of PIT565 and to identify maximal tolerated doses (MTDs) and/or recommended doses (RDs), schedule and route of administration in relapsed and/or refractory B-cell Non-Hodgkin lymphoma (R/R B-NHL) and relapsed and/or refractory B-cell acute lymphoblastic leukemia (R/R B-ALL).

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase I study of PIT565 in patients with R/R B-NHL and R/R B-ALL.

The study comprises a dose escalation part of PIT565 in two independent groups (group A: R/R B-NHL and B: R/R B-ALL) and a dose expansion part in three independent groups (R/R large B-cell lymphoma (LBCL) randomized in 1:1 ratio to two RDs (A1 and A2), and R/R B-ALL (B1)).

During the dose escalation, the safety (including the dose-dose limiting toxicity (DLT) relationship) and tolerability of PIT565 will be assessed, and schedule(s), route(s) of administration and dose(s) will be identified for use in the expansion part based on the review of these data. The RD will also be guided by the available information on pharmacokinetics (PK), pharmacodynamics (PD), and preliminary anti-tumor activity. The dose escalation will be guided by an adaptive Bayesian logistic regression model (BLRM) following the Escalation with Overdose Control (EWOC) principle.

Different schedules and routes of administrations will be explored in the dose escalation groups.

The dose expansion will further explore the MTD(s) and/or RD(s) and the selected schedule(s) and route of administration(s) in the three patients' groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Male or female patients ≥18 years of age at the date of signing the informed consent form
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2

NHL patient population

* Refractory or relapsed B-NHL
* Must have relapsed after or failed to respond to at least two prior treatment therapies including an αCD20 monoclonal antibody containing chemotherapy combination regimen
* Must have at least one bi-dimensionally measurable nodal lesion or one bi-dimensionally measurable extranodal lesion, as measured on positron emission tomography-computed tomography (PET/CT) scan

ALL patient population

* Refractory or relapsed CD19-positive B-ALL
* Morphologic disease in the bone marrow (≥ 5% blasts)

Exclusion Criteria:

* History of severe hypersensitivity to any ingredient of the study treatment or its excipients
* Contraindication to tocilizumab
* History of ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection
* Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type
* Active central nervous system (CNS) involvement by malignancy or presence of symptomatic CNS metastases, or CNS metastases that require local CNS-directed therapy (such as radiotherapy or surgery), or increasing doses of corticosteroids within the 2 weeks prior to the start of study treatment
* Active, known or suspected autoimmune disease other than patients with vitiligo, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur
* Patients receiving systemic treatment with any immunosuppressive medication

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2027-06-07 (Estimated); Study Completion 2028-06-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Dose Limiting Toxicities (DLTs) | 28 days or 35 days, depending on the dosing schedule
  Assessment of safety of study drug. A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value of CTCAE grade 3 or higher that occurs within the DLT evaluation period (28 days or 35 days depending on the schedule) and that is not primarily related to disease, disease progression, intercurrent illness, or concomitant medications with exceptions provided in the clinical protocol.
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 21 months
  Assessment of safety of study drug.
Frequency of dose interruptions | 21 months
  Assessment of tolerability of study drug
Frequency of dose reductions | 21 months
  Assessment of tolerability of study drug
Dose intensities | 21 months
  Assessment of tolerability of study drug Dose intensity is defined as the ratio of actual cumulative dose received and actual duration of exposure.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 21 months
  Evaluation of anti-tumor activity of PIT565 for Non-Hodgkin Lymphoma will be based on the Lugano Response Criteria Classification and anti-tumor activity of PIT565 for Acute Lymphoblastic Leukemia will be based on National Comprehensive Cancer Network (NCCN) 2018 v1 guidelines. Local investigator assessment will be used for analysis of efficacy endpoints.
Complete Response (CR) rate | 21 months
  Evaluation of anti-tumor activity of PIT565 for Non-Hodgkin Lymphoma will be based on the Lugano Response Criteria Classification and anti-tumor activity of PIT565 for Acute Lymphoblastic Leukemia will be based on National Comprehensive Cancer Network (NCCN) 2018 v1 guidelines. Local investigator assessment will be used for analysis of efficacy endpoints.
Best Overall Response (BOR) | 21 months
  Evaluation of anti-tumor activity of PIT565 for Non-Hodgkin Lymphoma will be based on the Lugano Response Criteria Classification and anti-tumor activity of PIT565 for Acute Lymphoblastic Leukemia will be based on National Comprehensive Cancer Network (NCCN) 2018 v1 guidelines. Local investigator assessment will be used for analysis of efficacy endpoints.
Duration Of Response (DOR) | 21 months
  Evaluation of anti-tumor activity of PIT565 for Non-Hodgkin Lymphoma will be based on the Lugano Response Criteria Classification and anti-tumor activity of PIT565 for Acute Lymphoblastic Leukemia will be based on National Comprehensive Cancer Network (NCCN) 2018 v1 guidelines. Local investigator assessment will be used for analysis of efficacy endpoints.
Overall Survival (OS) | 33 months
  Evaluation of anti-tumor activity of PIT565 for Non-Hodgkin Lymphoma will be based on the Lugano Response Criteria Classification and anti-tumor activity of PIT565 for Acute Lymphoblastic Leukemia will be based on National Comprehensive Cancer Network (NCCN) 2018 v1 guidelines. Local investigator assessment will be used for analysis of efficacy endpoints.
Progression Free Survival (PFS) | 21 months
  Evaluation of anti-tumor activity of PIT565 for Non-Hodgkin Lymphoma will be based on the Lugano Response Criteria Classification Local investigator assessment will be used for analysis of efficacy endpoints.
Event-free survival (EFS) | 21 months
  Evaluation of anti-tumor activity of PIT565 for Acute Lymphoblastic Leukemia will be based on National Comprehensive Cancer Network (NCCN) 2018 v1 guidelines. Local investigator assessment will be used for analysis of efficacy endpoints.
Maximum concentration of PIT565 (Cmax) | 21 months
  Pharmacokinetics (PK) parameters will be determined using non-compartmental method(s)
Area Under the Curve of PIT565 (AUC) | 21 months
  Pharmacokinetics (PK) parameters will be determined using non-compartmental method(s)
Trough concentration of PIT565 (C trough) | 21 months
  Pharmacokinetics (PK) parameters will be determined using non-compartmental method(s)
Prevalence of Anti-drug antibodies (ADA) at baseline | Baseline
  Assessment of anti-PIT565 antibodies in serum.
Incidence of Anti-drug antibodies (ADA) on treatment | 21 months
  Assessment of anti-PIT565 antibodies in serum.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (5):
  - University Of Miami, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - The University of Kansas Clinical Research Ctr, Fairway, Kansas
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - Oregon Health Sciences University, Portland, Oregon
- Novartis Investigative Site, Ghent, Belgium
- China (3):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- France (2):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Marseille
- Novartis Investigative Site, Tel Aviv, Israel
- Italy (2):
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Reggio Emilia, RE
- Novartis Investigative Site, Kashiwa, Chiba, Japan
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona

IPD SHARING:
Plan to Share IPD: No